CLINICAL TRIAL: NCT03790475
Title: Participation In Competing Strategies for COLorectal Cancer screenINg - a randOmized Health Services Study Within the National Screening Program in Poland(PICCOLINO)
Brief Title: Participation in Competing Strategies for Colorectal Cancer Screening - a Randomized Health Services Study Within the National Screening Program in Poland
Acronym: PICCOLINO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Ministry of Health, Poland (Other Government); Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Michal F. Kaminski, MD, PhD, MD, PhD, Maria Sklodowska-Curie National Research Institute of Oncology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 43/PB/2018
Record Dates: First submitted 2018-12-21; First posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer Screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Current screening practice. (No Intervention): Subjects randomized into this group will receive named invitations for colonoscopy with pre-specified date, contact details of dedicated screening center. Invitations will be sent 6 weeks prior to suggested date of screening test. All subjects not responding to the invitation will receive a reminder letter 3 weeks prior to proposed appointment date. Additionally, a re-invitation for colonoscopy (screening test in 6 weeks) will be sent to participants not responding to the first invitation and the reminding letter.
- Sequential screening strategy. (Experimental): Subjects randomized into this group will be initially invited to participate in a screening colonoscopy as per group 1. All subjects who will refuse colonoscopy or do not respond to invitation within 6 weeks since the first letter, will receive another invitation letter with FIT test enclosed.
  The screening office will contact persons with a positive test result in order to determine the date of the colonoscopy appointment.
  A negative test result will be sent together with a recommendation to have another screening test performed 2 years later and information about the possible delivery of the test in two years.
  Interventions: Other: Offering an alternative colorectal cancer screening method
- Multiple options screening strategy. (Experimental): Subjects in this group will receive a letter with an offer to choose between colonoscopy or FIT screening.
  The first letter will include an invitation with a scheduled date of colonoscopy (in 6 weeks) and a FIT kit.
  Three weeks before a scheduled date of colonoscopy subjects randomized into this group will receive a reminder letter with an information about proposed screening methods. After the scheduled date of the colonoscopy examination, subjects who will not respond to the invitation for colonoscopy and will not send the FIT test back to the laboratory will receive another invitation for colonoscopy (in 6 weeks) and a FIT kit.
  Interventions: Other: Offering a choice for colorectal cancer screening

INTERVENTIONS:
Other: Offering a choice for colorectal cancer screening — Persons randomized to the multiple options screening strategy group will receive a postal invitation offering a choice between FIT and colonoscopy.
  Arms: Multiple options screening strategy.
Other: Offering an alternative colorectal cancer screening method — Persons randomized to the sequential screening strategy group will receive a postal invitation to the colonoscopy followed by a postal invitation for screening using FIT for non-responders and subjects refusing colonoscopy.
  Arms: Sequential screening strategy.

SUMMARY:
The PICCOLINO is a randomized health services study performed within the framework of the Polish Colonoscopy Screening Program (PCSP) in Poland.

Within the study 12,298 eligible persons between 55 and 64 years of age will be drawn from the Population Registry and randomly assigned in a 1:1:1 ratio to receive an invitation to participate in one of the three screening strategies: (I) postal invitation to colonoscopy and a re-invitation to colonoscopy for initial non-responders, (II) postal invitation for screening using fecal immunochemical test (FIT) for non-responders and subjects refusing a colonoscopy, or (III) postal invitation offering a choice between FIT and colonoscopy.

Colonoscopies will be performed in seven local centers participating in the study. FITs will be analyzed in the central laboratory. Subjects with positive FIT result will be recommended to undergo colonoscopy.

The primary outcome is participation with CRC screening within 18 weeks after enrollment, defined as completion of colonoscopy, or completion of FIT along with colonoscopy for positive FIT result. Secondary outcome will be diagnostic yield for advanced neoplasia (CRC or advanced adenoma). The study has been approved by a local bioethics committee.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 55 to 64 years residing in Poland and assigned to be invited to screening within the Polish Colonoscopy Screening Program .

Exclusion Criteria:

* information of a selected subject death informed by family, neighbors or post office that has not been included in the Personal Identity Number (PESEL) system.
* addressees of letters that have been returned by the post office.
* subjects requiring long-term care due to somatic, psychosocial reasons or with mental disability.
* history of colorectal resection.

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12298 (Estimated)
Dates: Start 2018-08-25 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Completion of the assigned screening strategy within 18 weeks of enrollment | Within 18 weeks of enrollment
  Completion of the assigned screening strategy within 18 weeks of enrollment defined as:
  * current screening strategy: documented screening colonoscopy,
  * sequential and multiple options strategies: documented colonoscopy, or receipt of FIT containing stool specimen. A positive FIT result requires subsequent documented colonoscopy to qualify as completed.

SECONDARY OUTCOMES:
Diagnostic yield for CRC and advanced adenomas | Within 18 weeks of enrollment
  Advanced adenoma defined as adenoma >1 cm in size, or with high-grade dysplasia, or with villous component (>25%).

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Sklodowska-Curie Institute - Oncology Center, Warsaw, Poland

REFERENCES:
- [Derived] Pilonis ND, Bugajski M, Wieszczy P, Rupinski M, Pisera M, Pawlak E, Regula J, Kaminski MF. Participation in Competing Strategies for Colorectal Cancer Screening: A Randomized Health Services Study (PICCOLINO Study). Gastroenterology. 2021 Mar;160(4):1097-1105. doi: 10.1053/j.gastro.2020.11.049. Epub 2020 Dec 9. PMID 33307024